CLINICAL TRIAL: NCT01571206
Title: An Open-Label, Single-Arm, Extension Study to Demonstrate Long-Term Efficacy and Safety of CT-P13 in Patients With Ankylosing Spondylitis Who Were Treated With Infliximab (Remicade or CT-P13) in Study CT-P13 1.1
Brief Title: An Extension Study to Demonstrate the Equivalence of Long-Term Efficacy and Safety of CT-P13 in Patients With Ankylosing Spondylitis Who Were Treated With Infliximab (Remicade or CT-P13) in Study CT-P13 1.1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-P13 1.3; 2011-004572-11 (EudraCT Number)
Record Dates: First submitted 2012-03-23; First posted 2012-04-05 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Ankylosing Spondylitis
Keywords: AS; Biosimilar
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CT-P13 (Active Comparator): infliximab
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — CT-P13 (5mg/kg) administered as a 2-hour IV infusion per dose

SUMMARY:
This open-label, single-arm, multicenter, multiple single-dose intravenous (IV) infusion, efficacy, and safety extension study of the Phase 1 Study CT-P13 1.1 is designed to assess the long-term efficacy and safety of multiple doses of CT-P13.

ELIGIBILITY:
Inclusion Criteria:

* Patient who has completed the scheduled visits, including the End-of-Study Visit, in Study CT-P13 1.1
* Patient who has not had any major protocol violation in Study CT-P13 1.1

Exclusion Criteria:

* Patient who has been withdrawn from Study CT-P13 1.1 for any reason
* Patient who, at the time of providing informed consent, has any ongoing medical issues such as serious adverse events(SAEs) or intolerance issues that mean continuation in this extension study could be detrimental to their health, in the option of the investigator
* Patient who plans to participate in a study with an investigational drug during the period of this extension study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Long term efficacy evaluated by Assessment of Spondylo Arthritis International Society(ASAS) criteria and Long term safety evaluated by immunogenicity and clinical laboratory test | Up to Week 40

CONTACTS AND LOCATIONS:
Overall Officials: Won Park, M.D., Ph.D., Study Director — Inha University Hospital
Locations (1):
- Inha University Hospital, Incheon, South Korea

REFERENCES:
- [Derived] Park W, Yoo DH, Miranda P, Brzosko M, Wiland P, Gutierrez-Urena S, Mikazane H, Lee YA, Smiyan S, Lim MJ, Kadinov V, Abud-Mendoza C, Kim H, Lee SJ, Bae Y, Kim S, Braun J. Efficacy and safety of switching from reference infliximab to CT-P13 compared with maintenance of CT-P13 in ankylosing spondylitis: 102-week data from the PLANETAS extension study. Ann Rheum Dis. 2017 Feb;76(2):346-354. doi: 10.1136/annrheumdis-2015-208783. Epub 2016 Apr 26. PMID 27117698